CLINICAL TRIAL: NCT02453477
Title: A Phase I/II Study Evaluating Safety and Efficacy of Autologous Hematopoietic Stem Cells Genetically Modified With GLOBE Lentiviral Vector Encoding for the Human Beta-globin Gene for the Treatment of Patients Affected by Transfusion Dependent Beta-thalassemia
Brief Title: Gene Therapy for Transfusion Dependent Beta-thalassemia
Acronym: TIGET-BTHAL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Fondazione Telethon (Other); Orchard Therapeutics (Industry)
Responsible Party: Principal Investigator, Alessandro Aiuti, Director of Pediatric Clinical Research Unit, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-004860-39 (EudraCT)
Record Dates: First submitted 2015-05-15; First posted 2015-05-25 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Beta-Thalassemia
Keywords: Beta thalassemia; Gene therapy; Lentiviral vector
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Adults (Experimental): ≥18 years (3 subjects) The ATIMP consists of autologous CD34+ cell enriched fraction containing hematopoietic stem cells (HSC) transduced with the GLOBE lentiviral vector encoding for the beta-globin gene re-suspended in their final formulation medium.
  Dosage indications The target dose in the transduced product is 5x10(6) cells/Kg CD34+cells, with a minimum dose of 2x10(6)/Kg and a maximum dose of 20x10(6)/Kg, depending on the yield of cells.
  The product will be injected intraosseously.
  Interventions: Genetic: Autologous hematopoietic stem cells genetically modified with GLOBE lentiviral vector encoding for the human beta-globin gene
- Elderly children (Experimental): 8-17 years (3 subjects) The ATIMP consists of autologous CD34+ cell enriched fraction containing hematopoietic stem cells (HSC) transduced with the GLOBE lentiviral vector encoding for the beta-globin gene re-suspended in their final formulation medium.
  Dosage indications The target dose in the transduced product is 5x10(6) cells/Kg CD34+cells, with a minimum dose of 2x10(6)/Kg and a maximum dose of 20x10(6)/Kg, depending on the yield of cells.
  The product will be injected intraosseously.
  Interventions: Genetic: Autologous hematopoietic stem cells genetically modified with GLOBE lentiviral vector encoding for the human beta-globin gene
- Younger children (Experimental): 3-7 years (4 subjects) The ATIMP consists of autologous CD34+ cell enriched fraction containing hematopoietic stem cells (HSC) transduced with the GLOBE lentiviral vector encoding for the beta-globin gene re-suspended in their final formulation medium.
  Dosage indications The target dose in the transduced product is 5x10(6) cells/Kg CD34+cells, with a minimum dose of 2x10(6)/Kg and a maximum dose of 20x10(6)/Kg, depending on the yield of cells.
  The product will be injected intraosseously.
  Interventions: Genetic: Autologous hematopoietic stem cells genetically modified with GLOBE lentiviral vector encoding for the human beta-globin gene

INTERVENTIONS:
Genetic: Autologous hematopoietic stem cells genetically modified with GLOBE lentiviral vector encoding for the human beta-globin gene — Autologous CD34+ cell enriched fraction containing hematopoietic stem cells (HSC) transduced with the GLOBE lentiviral vector encoding for the human beta-globin gene resuspended in their final formulation medium. The target dose in the transduced product is 5x10^6 cells/Kg CD34+ cells, with a minimum dose of 2 x 10^6/Kg and a maximum dose of 20 x 10^6/Kg, depending on the yield of cells. The product will be injected intraosseously.

SUMMARY:
This is a phase I/II study evaluating safety and efficacy of autologous hematopoietic stem cells genetically modified with GLOBE lentiviral vector encoding for the human beta-globin gene for the treatment of patients affected by transfusion dependent beta-thalassemia

DETAILED DESCRIPTION:
Both adults and pediatric patients will be treated with genetically modified autologous hematopoietic stem cells collected from mobilized peripheral blood (or bone marrow for patients < 8 years in case mobilization will not be feasible) and transduced with GLOBE lentiviral vector encoding for the human beta-globin gene.

This study will enroll 10 patients allocated in 3 groups, according to age and conditioning regimen:

1. 3 adults (≥18 years) conditioned with treosulfan and thiotepa
2. 3 elderly children (8-17 years) conditioned with treosulfan and thiotepa
3. 4 younger children (3-7 years) conditioned with treosulfan and thiotepa Enrolment will start in adult patients. Pediatric patients will be included once evidence of preliminary safety and biological efficacy is shown in at least 2 adults.

Patients are included regardless of the beta globin gene mutation, provided an adequate cardiac, renal, hepatic and pulmonary function is demonstrated. Patients with severe iron overload are excluded as well as patients with active viral infections. Pediatric patients can be enrolled only in absence of a human leukocyte antigen (HLA)-identical sibling or a suitable 10/10 matched unrelated donor.

The treated patients will be followed for 2 years. After completion of the 2 years follow up, patients will be enrolled in a long term follow up study and followed up for at least other additional 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Transfusion-dependent beta-thalassemia (any genotype). Transfusion dependence is defined as receiving ≥ 8 transfusions of blood per year over a minimum of 2 years.
* Karnofsky Index or Lansky > 80%
* Age ≥ 3 years and < 65 years
* Adequate cardiac, renal, hepatic and pulmonary functions as evidenced by:

  * Left ventricular ejection fraction (LVEF) greater than 45% by echo and normal ECG or presence of abnormalities not significant for cardiac disease. Absence of severe pulmonary hypertension
  * Diffusing capacity of the lung for carbon monoxide (DLCO) > 50% and forced expiratory volume in 1 sec (FEV1) and forced expiratory vital capacity (FVC) > 60% predicted (if non cooperative: pulse oximetry > 95 % in room air)
  * Serum creatinine < 1.5 upper limit of normal
  * Absent-mild-moderate liver iron overload on T2*MRI (less than 12 months before enrolment)
  * Absent-mild-moderate cardiac iron overload T2*MRI (less than 12 months before enrolment)
  * Absence of severe liver fibrosis or cirrhosis on fibroscan or liver biopsy (less than 12 months before enrolment)
* Low risk thrombophilic screen and negative history of significant previous thrombotic events
* For all patients in reproductive age, agreement to use highly effective and adequate method of contraception while receiving treatment phase and for at least 12 months following drugs administration (including both females of child bearing potential and males with partners of child bearing potential)
* Good adherence to transfusion and chelation programme as indirect evidence of good adherence to treatment and follow-up evaluations for current trial
* Availability of an adequate and well documented transfusion history (at least previous 6 months) or availability to follow a regular transfusion regimen according to guidelines and provide a detailed transfusion record of the 6 months prior to intervention phase

Exclusion Criteria:

* Use of other investigational agents within 4 weeks prior to study enrolment (within 6 weeks if use of long-acting agents)
* Severe, active viral, bacterial, or fungal infection at eligibility evaluation
* Malignant neoplasia (except local skin cancer or cervical intraepithelial neoplasia) or exceptional family history of familial cancer syndromes
* Myelodysplasia, cytogenetic alterations associated with neoplasia, or other serious haematological disorder than thalassemia
* History of uncontrolled seizures
* Other clinical conditions judged non compatible with the procedure and/or the treatment
* Positivity for HIV (serology or RNA), and/or HbsAg and/or HBV DNA and/or HCV RNA (or negative HCV RNA but on antiviral treatment) and/or Treponema Pallidum or Mycoplasma active infection
* Active alcohol or substance abuse within 6 months of the study
* Pregnancy or lactation
* Previous allogeneic bone marrow transplantation or gene therapy
* For paediatric patients only: availability of an HLA-matched donor (sibling or of a suitable 10/10 matched unrelated donor).

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Number of patients alive all over the trial
Achievement of hematological engraftment | within day +60 after gene therapy
  Haematological engraftment is defined as first day of neutrophil count >500/mm3 and platelets >20,000/mm3 on 3 consecutive blood counts.
Safety of the administration of autologous haematopoietic stem cells transduced with LV-GLOBE | 0-24 months after gene therapy
  * short-term tolerability: the percentage of patients not experiencing short-term (0-24 hours from injection) adverse events (of any grade) and systemic reactions.
  * absence of Replication Competent Lentivirus (RCL): the percentage of subjects without RCL in the 24 months from injection.
  * absence of abnormal clonal proliferation: the percentage of subjects without abnormal clonal proliferation in the 24 months from injection.
Short-term safety and tolerability of the different conditioning regimens | from day -5 (first day of conditioning treatment) to day 100 after gene therapy
  The percentage of patients with the following clinical events from day -5 to +100 days from injection: NCI (National Cancer Institute Common Terminology Criteria grading) ≥2 and metabolic/laboratory NCI ≥3.
Overall safety and tolerability measured by AE recording | 0-24 months after gene therapy
  The number of AEs (adverse events) and SAEs (serious adverse events) and the percentage of subjects experiencing AEs and SAEs in the 24 months post injection will be summarized by severity and within body system involved.
Polyclonal engraftment | From 6 months to 2 years after gene therapy
  The percentage of subjects with polyclonality of haematopoiesis will be estimated at 6, 12, 18 and 24 months from injection. Polyclonality of haematopoiesis will be defined as > 1000 unique integration sites retrieved from peripheral blood and/or bone marrow cells.
Reduction in transfusion frequency up to transfusion independence | from -7 months before gene therapy to 2 years after gene therapy
  Transfusions will be recorded as mLs of blood/kg/months

SECONDARY OUTCOMES:
Transfusion independence | 9 months, 1, 1.5 and 2 years after gene therapy
  Transfusion independence is defined as ≤ 1 transfusion in the previous 6 months
Adequate haemoglobin level | 0-24 months after gene therapy
  Haemoglobin level will be assessed by full blood counts in patients achieving transfusion independence. Adequate haemoglobin is defined as haemoglobin >9 g/dl in adults and >10 g/dl in children.
Adequate engraftment of genetically corrected cells | 6, 12, and 24 months after gene therapy
  Engraftment will be assessed by vector-specific quantitative Polymerase Chain reaction (PCR) on bone marrow. Adequate engraftment is defined as ≥ 0.15 VCN/genome. (VCN = Vector Copy Number)
Transgene expression | 6, 12, and 24 months after gene therapy
  Transgene expression will be evaluated by globin chains and/or hemoglobin synthesis on peripheral blood and/or bone marrow samples by HPLC and/or electrophoresis analysis
Improvement of health-related quality of life | 12 and 24 months
  Health-related quality of life will be assessed by the use of standardized questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Aiuti, MD, PhD, Principal Investigator — Ospedale San Raffaele; Fabio Ciceri, MD, Study Chair — Ospedale San Raffaele; Sarah Marktel, MD, Study Chair — Ospedale San Raffaele; Maria Domenica Cappellini, MD, Study Chair — IRCCS Policlinico Foundation; Giuliana Ferrari, PhD, Study Director — Telethon Institute of Gene Therapy, Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Background] Aiuti A, Biasco L, Scaramuzza S, Ferrua F, Cicalese MP, Baricordi C, Dionisio F, Calabria A, Giannelli S, Castiello MC, Bosticardo M, Evangelio C, Assanelli A, Casiraghi M, Di Nunzio S, Callegaro L, Benati C, Rizzardi P, Pellin D, Di Serio C, Schmidt M, Von Kalle C, Gardner J, Mehta N, Neduva V, Dow DJ, Galy A, Miniero R, Finocchi A, Metin A, Banerjee PP, Orange JS, Galimberti S, Valsecchi MG, Biffi A, Montini E, Villa A, Ciceri F, Roncarolo MG, Naldini L. Lentiviral hematopoietic stem cell gene therapy in patients with Wiskott-Aldrich syndrome. Science. 2013 Aug 23;341(6148):1233151. doi: 10.1126/science.1233151. Epub 2013 Jul 11. PMID 23845947
- [Background] Aiuti A, Cassani B, Andolfi G, Mirolo M, Biasco L, Recchia A, Urbinati F, Valacca C, Scaramuzza S, Aker M, Slavin S, Cazzola M, Sartori D, Ambrosi A, Di Serio C, Roncarolo MG, Mavilio F, Bordignon C. Multilineage hematopoietic reconstitution without clonal selection in ADA-SCID patients treated with stem cell gene therapy. J Clin Invest. 2007 Aug;117(8):2233-40. doi: 10.1172/JCI31666. PMID 17671653
- [Background] Aiuti A, Cattaneo F, Galimberti S, Benninghoff U, Cassani B, Callegaro L, Scaramuzza S, Andolfi G, Mirolo M, Brigida I, Tabucchi A, Carlucci F, Eibl M, Aker M, Slavin S, Al-Mousa H, Al Ghonaium A, Ferster A, Duppenthaler A, Notarangelo L, Wintergerst U, Buckley RH, Bregni M, Marktel S, Valsecchi MG, Rossi P, Ciceri F, Miniero R, Bordignon C, Roncarolo MG. Gene therapy for immunodeficiency due to adenosine deaminase deficiency. N Engl J Med. 2009 Jan 29;360(5):447-58. doi: 10.1056/NEJMoa0805817. PMID 19179314
- [Background] Biffi A, Montini E, Lorioli L, Cesani M, Fumagalli F, Plati T, Baldoli C, Martino S, Calabria A, Canale S, Benedicenti F, Vallanti G, Biasco L, Leo S, Kabbara N, Zanetti G, Rizzo WB, Mehta NA, Cicalese MP, Casiraghi M, Boelens JJ, Del Carro U, Dow DJ, Schmidt M, Assanelli A, Neduva V, Di Serio C, Stupka E, Gardner J, von Kalle C, Bordignon C, Ciceri F, Rovelli A, Roncarolo MG, Aiuti A, Sessa M, Naldini L. Lentiviral hematopoietic stem cell gene therapy benefits metachromatic leukodystrophy. Science. 2013 Aug 23;341(6148):1233158. doi: 10.1126/science.1233158. Epub 2013 Jul 11. PMID 23845948
- [Background] Frittoli MC, Biral E, Cappelli B, Zambelli M, Roncarolo MG, Ferrari G, Ciceri F, Marktel S. Bone marrow as a source of hematopoietic stem cells for human gene therapy of beta-thalassemia. Hum Gene Ther. 2011 Apr;22(4):507-13. doi: 10.1089/hum.2010.045. Epub 2011 Mar 4. PMID 20979441
- [Background] Miccio A, Cesari R, Lotti F, Rossi C, Sanvito F, Ponzoni M, Routledge SJ, Chow CM, Antoniou MN, Ferrari G. In vivo selection of genetically modified erythroblastic progenitors leads to long-term correction of beta-thalassemia. Proc Natl Acad Sci U S A. 2008 Jul 29;105(30):10547-52. doi: 10.1073/pnas.0711666105. Epub 2008 Jul 23. PMID 18650378
- [Background] Montini E, Cesana D, Schmidt M, Sanvito F, Ponzoni M, Bartholomae C, Sergi Sergi L, Benedicenti F, Ambrosi A, Di Serio C, Doglioni C, von Kalle C, Naldini L. Hematopoietic stem cell gene transfer in a tumor-prone mouse model uncovers low genotoxicity of lentiviral vector integration. Nat Biotechnol. 2006 Jun;24(6):687-96. doi: 10.1038/nbt1216. Epub 2006 May 28. PMID 16732270
- [Background] Roselli EA, Mezzadra R, Frittoli MC, Maruggi G, Biral E, Mavilio F, Mastropietro F, Amato A, Tonon G, Refaldi C, Cappellini MD, Andreani M, Lucarelli G, Roncarolo MG, Marktel S, Ferrari G. Correction of beta-thalassemia major by gene transfer in haematopoietic progenitors of pediatric patients. EMBO Mol Med. 2010 Aug;2(8):315-28. doi: 10.1002/emmm.201000083. PMID 20665635